CLINICAL TRIAL: NCT04848987
Title: Indirect Resin Composite Inlays Cemented With Three Different Luting Strategies
Brief Title: Indirect Resin Composite Inlays Cemented With a Self-adhesive, Self-etch or a Conventional Resin Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A10150421
Record Dates: First submitted 2021-04-10; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Dental Leakage
Keywords: Resin Composite; Randomized Clinical Trial; Operative Dentistry
MeSH Terms: conditions — Dental Leakage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Etch-and-rinse (Variolink N) resin cement (Active Comparator): For etch-and-rinse resin cement, 40 inlays were cemented by Variolink N resin cement.
  Interventions: Procedure: Etching
- Self-etch (Panavia F2.0) resin cement (Placebo Comparator): Regarding self-etch resin cement, 40 inlays were cemented by Panavia F2.0 resin cement.
  Interventions: Procedure: Etching
- Self-adhesive (RelyX Unicem) resin cement (No Intervention): For self-adhesive resin cement, 40 inlays were cemented by RelyX Unicem resin cement.

INTERVENTIONS:
Procedure: Etching — Etching enamel surface using phosphoric acid
  Arms: Etch-and-rinse (Variolink N) resin cement; Self-etch (Panavia F2.0) resin cement

SUMMARY:
The present study was designed to provide further evidence in this particular research prospective, and this study hence aimed to clinically evaluate the 5-years adhesion durability of indirect resin composite inlays luted with three different resin cement strategies in MOD Class II restorations. The formulated null hypothesis was that there is no significant difference in the clinical performances of the three different resin cement strategies for luting indirect resin composite inlays in MOD Class II restorations for 5-years.

The research question was as follows: Do self-adhesive resin cements in class II restorations present better clinical performances than conventional etch-and-rinse and self-etch resin cements according to the USPHS criteria?

DETAILED DESCRIPTION:
Objective: To clinically evaluate the 5 years adhesion durability of indirect resin composite inlays luted with three different resin cement strategies in MOD Class II restorations.

Materials and Methods: A randomized clinical trial was conducted following the protocol, 40 patients with three large cavities for each one that indicated for indirect MOD Class II restorations were enrolled in the current study. Then, 120 indirect resin composite inlay restorations (SR Nexco) were placed and luted with three different resin cement strategies; an etch-and-rinse (Variolink N), self-etch (Panavia F2.0) and self-adhesive (RelyX Unicem). Each resin cement was used for luting 20 inlay restorations. A single operator placed all restorations according to the manufacturer's instructions. Immediatelly after placement, the restorations were finished and polished. Clinical evaluation was performed at baseline and at 1, 3 and 5 years intervals after placement by two independent examiners using modified USPHS criteria. The changes in the USPHS parameters during the 5 years period were analyzed with Fredman test. The baseline scores were compared with those at the recall visits using Wilcoxon signed rank test, where the level of significance was set at p˂0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary caries involving occlusal surface only with ICDAS 2 and 3.
* Patients with cavities no more than one-third of the intercuspal distance.
* Patients must have a good oral hygiene.
* Patients with tooth gives positive response to testing with an electric pulp tester.
* Patients with normal and full occlusion.
* Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

* High caries risk patients with extremely poor oral hygiene.
* Patients involved in orthodontic treatment or periodontal surgery.
* Patients with periodontally involved teeth (chronic periodontitis).
* Patients with abutments should be excluded.
* Patients with heavy bruxism habits and clenching.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Percentage % of patients with marginal staining | 5 years after restoration procedure
  Percentage of marginal staining in patients was clinically assessed using USPHS criteria. Restorations were given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study Protocol, Statistical Analysis Plan can be shared to other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 3 Months for 5 years
Access Criteria: For anyone